CLINICAL TRIAL: NCT04660890
Title: A Multiple-Ascending-Dose, Randomized, Double-Blind, Double-Dummy, Placebo- and Positive-Controlled Study to Evaluate the Effect of ALXN2050 on the QT Interval in Healthy Adult Participants
Brief Title: A Study of the Cardiac Effects of ALXN2050 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ALXN2050-HV-107
Record Dates: First submitted 2020-11-12; First posted 2020-12-09 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-11

CONDITIONS: Healthy
Keywords: ALXN2050; Electrocardiogram; QT Interval; Concentration-QT; Factor D Inhibitor
MeSH Terms: interventions — rhoA GTP-Binding Protein; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Arm (ABC) (Experimental): Treatment Sequence ABC - Participants will receive all 3 doses of ALXN2050 in a multiple-ascending fashion over 3 periods:
  Treatment A (Period 1): ALXN2050 Dose 120 milligrams (mg) and moxifloxacin-matching placebo.
  Treatment B (Period 2): ALXN2050 Dose 240 mg and moxifloxacin-matching placebo.
  Treatment C (Period 3): ALXN2050 Dose 360 mg and moxifloxacin-matching placebo.
  Interventions: Drug: ALXN2050; Drug: Moxifloxacin-matching Placebo
- Control Arm (DEF) (Placebo Comparator): Treatment Sequence DEF - Participants will receive ALXN2050-matching placebo over 3 periods:
  Treatment D (Period 1): 120 mg ALXN2050-matching placebo and moxifloxacin-matching placebo.
  Treatment E (Period 2): 240 mg ALXN2050-matching placebo and moxifloxacin.
  Treatment F (Period 3): 360 mg ALXN2050-matching placebo and moxifloxacin-matching placebo.
  Interventions: Drug: ALXN2050-matching Placebo; Drug: Moxifloxacin; Drug: Moxifloxacin-matching Placebo
- Control Arm (GHI) (Placebo Comparator): Treatment Sequence GHI - Participants will receive ALXN2050-matching placebo over 3 periods:
  Treatment G (Period 1): 120 mg ALXN2050-matching placebo and moxifloxacin.
  Treatment H (Period 2): 240 mg ALXN2050-matching placebo and moxifloxacin-matching placebo.
  Treatment I (Period 3): 360 mg ALXN2050-matching placebo and moxifloxacin.
  Interventions: Drug: ALXN2050-matching Placebo; Drug: Moxifloxacin; Drug: Moxifloxacin-matching Placebo

INTERVENTIONS:
Drug: ALXN2050 — ALXN2050 will be administered orally twice daily as powder-in-capsule.
  Other Names: ACH-0145228 (formerly)
  Arms: Treatment Arm (ABC)
Drug: ALXN2050-matching Placebo — ALXN2050-matching placebo will be administered orally twice daily as placebo powder-in-capsule.
  Arms: Control Arm (DEF); Control Arm (GHI)
Drug: Moxifloxacin — Moxifloxacin will be administered as a single oral dose.
  Arms: Control Arm (DEF); Control Arm (GHI)
Drug: Moxifloxacin-matching Placebo — Moxifloxacin-matching placebo will be administered as a single oral dose.

SUMMARY:
This is a randomized, double-blind, double-dummy, placebo- and positive-controlled parallel study to evaluate the effect of ALXN2050 on the QT interval in healthy adult participants.

DETAILED DESCRIPTION:
Participants randomized to the treatment arm will receive ALXN2050 in a multiple-ascending doses fashion over 3 periods (treatment sequence ABC). Participants randomized to the control arms will be further randomized to 1 of 2 treatment sequences (treatment sequence DEF or GHI) to receive placebo or active control over 3 periods.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index in the range of 18.0 to 32.0 kilograms (kg)/meter squared, inclusive, with a minimum body weight of 50.0 kg at screening.
2. No clinically significant history or presence of ECG abnormalities at screening.
3. Female participants must be of non-childbearing potential and need not employ a method of contraception.
4. Non-sterile male participants must agree to abstinence or use a highly effective method of contraception.

Exclusion Criteria:

1. Clinically significant laboratory abnormalities.
2. History of any medical or psychiatric condition or disease that might limit the participant's ability to complete or participate in this clinical study, confound the results of the study, or pose an additional risk to the participant by their participation in the study.
3. History or presence of drug or alcohol abuse within previous 2 years, current tobacco and/or nicotine user, or positive alcohol and/or drug screen at screening or Day -1 of Period 1.
4. History or presence of clinically significant seizures, head injury, or head trauma.
5. History of procedures that could alter absorption or excretion of orally administered drugs.
6. History of meningococcal infection, or a first-degree relative with a history of meningococcal infection.
7. History of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs.
8. Body temperature ≥ 38.0°Celsius at screening or prior to first dosing in Period 1 or history of febrile illness, or other evidence of infection, within 14 days prior to (first) dosing.
9. Donation of whole blood from 3 months prior to first dosing, or of plasma from 30 days before first dosing, or receipt of blood products within 6 months prior to first dosing.
10. Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives (if known) or 30 days before first dosing, whichever is longer.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Placebo-corrected Change From Baseline QTc Intervals (ddQTc) For ALXN2050 | Pre-dose through 24 hours post-dose
  Twelve-lead electrocardiograms (ECGs) will be extracted from continuous (Holter) recordings.

SECONDARY OUTCOMES:
Change From Baseline PR Interval (dPR) For ALXN2050 | Pre-dose through 24 hours post-dose
  Twelve-lead ECGs will be extracted from continuous (Holter) recordings.
ddQTc For Moxifloxacin | Pre-dose through 24 hours post-dose
  Twelve-lead ECGs will be extracted from continuous (Holter) recordings.
Area Under The Plasma Concentration-time Curve During A Dosing Interval (tau) At Steady-state (AUCtau) For ALXN2050 | Pre-dose through 24 hours post-dose
Maximum Observed Plasma Concentration Following Multiple Dosing (Cmax,ss) For ALXN2050 | Up to 24 hours postdose
Time To Maximum Observed Plasma Concentration Following Multiple Dosing (Tmax,ss) For ALXN2050 | Pre-dose through 24 hours post-dose
Incidence Of Treatment-emergent Adverse Events | Day 1 (postdose) through follow-up (7 [+/- 2] days after last study drug administration)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No